CLINICAL TRIAL: NCT05865210
Title: Effects of Kegel Exercises With and Without Myofascial Release on Pain, Function and Quality of Life in Chronic Pelvic Pain
Brief Title: Effects of Kegel Exercises With and Without Myofascial Release in Chronic Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0525
Record Dates: First submitted 2023-04-18; First posted 2023-05-18 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Chronic Pelvic Pain Syndrome
MeSH Terms: interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kegel Exercise with Myofascial release technique group: (Experimental): Group A, we told patient to perform kegel exercise by hold and relax the pelvic floor muscles, initially 3-4 contractions for 3-5 seconds then we increase the repetition according to patient and apply myofascial release for trigger points. 4 session per week and post intervention assessment after 3 weeks follow-up
  Interventions: Other: Kegel Exercise; Other: Myofascial release technique
- Kegel Exercise group (Active Comparator): Group B, In this group we only perform kegel exercises to patients as hold and relax of pelvic floor muscle 3-4 contraction for 3-5 seconds.4 session per week and post intervention assessment after 3 weeks follow-up
  Interventions: Other: Kegel Exercise

INTERVENTIONS:
Other: Kegel Exercise — Kegel exercises (also called pelvic floor exercises) will be used to strengthen the pelvic floor muscles it will involve repeatedly contracting and relaxing the muscles that form part of the pelvic floor.
Other: Myofascial release technique — Myofasical release will include deep pressure for 10-15 seconds to release the trigger points and also gentle, light soft tissue massage on the vaginal muscles and surrounding areas.
  Arms: Kegel Exercise with Myofascial release technique group:

SUMMARY:
Study will be a Randomized control trial to check the effects of kegel exercise with and without myofascial release on chronic pelvic pain in females so that we can examine the effect of above techniques on pain, function and quality of life in chronic pelvic pain females.Non-probability convenience sampling technique will be used, subject following eligibility criteria from DHQ Hospital Layyah will be randomly allocated in two groups. Group A participants will be given kegel exercise with myofascial release, Group B participants will be given kegel exercise for 3 weeks. Assessment will be done via, Numeric Pain Rating Scale and pelvic floor impact questionnaire (PFIQ) and functional pelvic pain scale

DETAILED DESCRIPTION:
Chronic pelvic pain (CPP), defined as a noncyclical pain lasting for more than 6 months can lead to lower physical performance and quality of life in women. In this study the effects of Kegel Exercise with and without myofascial release in chronic pelvic pain population will be analyzed. This study will be a randomized clinical trial. Kegel Exercise and Myofasical Release would be administered to the chronic Pelvic pain Females. Subjects meeting the predetermined inclusion criteria will be divided into two groups. Assessment will be done using Numeric Pain rating scale (NPR), Pelvic floor Impact Questionnaire (PFIQ) and Functional pelvic pain scale (FPPS). Subjects in one group will be treated with kegel exercise with myofascial release, and the other will be treated with kegel exercise only. Each subject will receive a total 12 treatment sessions, with 04 treatment sessions per week. Measurements will be recorded at start and end of treatment session. Recorded values will be analyzed for any change using SPSS.

ELIGIBILITY:
Inclusion Criteria:

* • Age 25-55

  * Record of CPPS for more than 6 months.
  * Complete gynaecological consultation with necessary workup.
  * Chronic pelvic pain associated with gynaecological issue.
  * Patients who have tenderness upon palpation are included, suggesting that the trigger points are painful.
  * Patient that can't cope with their daily activities

Exclusion Criteria:

* Acute active infection
* Malignancy
* Active pregnancy
* Pudendal nerve entrapment syndrome.
* Not simultaneously partaking in pelvic floor physical therapy.
* No evoked tenderness upon palpation of levator ani sling at examination.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 3 weeks
  The NPRS is a segmented numeric scale in which the respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. NPRS is anchored by terms describing pain severity extremes. changes from Baseline to 3 week
Pelvic floor Impact Questionnaire (PFIQ): | 3 weeks
  The PFIQ-7 consists of 7 questions that need to be answered 3 times each (corresponds to the scales previously mentioned) considering symptoms related to the bladder or urine, vagina or pelvis, and bowel or rectum and their effect on function, social health, and mental health in the past 3 months. The scale scores are then added together to get the total PFIQ-7 score, which ranges from 0-300. A lower score means there is a lesser effect on quality of life. changes from Baseline to 3 week
Functional pelvic pain scale: | 3 weeks
  The FPPS is a sensitive and reliable measure of pelvic pain intensity through, time, demonstrating evidence of validity. Functional Pelvic Pain Scale (FPPS), designed to measure pelvic pain intensity as it relates to functions of daily living (bladder and bowel function, intercourse, walking, running, lifting, working, and sleeping). changes from Baseline to 3 week

CONTACTS AND LOCATIONS:
Overall Officials: Tooba Zahid, MS*, Principal Investigator — Riphah International University
Locations (1):
- District Headquarters Hospital, Layyah, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrews J, Yunker A, Reynolds WS, Likis FE, Sathe NA, Jerome RN. Noncyclic Chronic Pelvic Pain Therapies for Women: Comparative Effectiveness [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2012 Jan. Report No.: 11(12)-EHC088-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK84586/ PMID 22439157
- [Background] Ahangari A. Prevalence of chronic pelvic pain among women: an updated review. Pain Physician. 2014 Mar-Apr;17(2):E141-7. PMID 24658485
- [Background] Fillingim RB, King CD, Ribeiro-Dasilva MC, Rahim-Williams B, Riley JL 3rd. Sex, gender, and pain: a review of recent clinical and experimental findings. J Pain. 2009 May;10(5):447-85. doi: 10.1016/j.jpain.2008.12.001. PMID 19411059
- [Background] Unruh AM. Gender variations in clinical pain experience. Pain. 1996 May-Jun;65(2-3):123-67. doi: 10.1016/0304-3959(95)00214-6. PMID 8826503
- [Background] Wiesenfeld-Hallin Z. Sex differences in pain perception. Gend Med. 2005 Sep;2(3):137-45. doi: 10.1016/s1550-8579(05)80042-7. PMID 16290886
- [Background] Giamberardino MA. Women and visceral pain: are the reproductive organs the main protagonists? Mini-review at the occasion of the "European Week Against Pain in Women 2007". Eur J Pain. 2008 Apr;12(3):257-60. doi: 10.1016/j.ejpain.2007.11.007. Epub 2008 Jan 14. No abstract available. PMID 18249016
- [Background] Harlow BL, Stewart EG. A population-based assessment of chronic unexplained vulvar pain: have we underestimated the prevalence of vulvodynia? J Am Med Womens Assoc (1972). 2003 Spring;58(2):82-8. PMID 12744420
- [Background] Wu WH, Meijer OG, Uegaki K, Mens JM, van Dieen JH, Wuisman PI, Ostgaard HC. Pregnancy-related pelvic girdle pain (PPP), I: Terminology, clinical presentation, and prevalence. Eur Spine J. 2004 Nov;13(7):575-89. doi: 10.1007/s00586-003-0615-y. Epub 2004 Aug 27. PMID 15338362